CLINICAL TRIAL: NCT00207896
Title: Defining the Prevalence of Acute Neuroendocrine Dysfunction and Correlating the Dysfunction With Outcomes in Critically Ill Pediatric Patients: A Pilot Study
Brief Title: Neuroendocrine Dysfunction in Critically Ill Pediatric Patients
Status: Completed | Type: Observational
Sponsor: Children's Healthcare of Atlanta (Other)
Responsible Party: Sponsor
Other Study IDs: 04-068
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Critical Illness
Keywords: Pediatric Intensive Care; Neuroendocrine Dysfunction
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Research studies in adults have shown that certain hormones may be decreased or may not work normally which contributes to how sick a person becomes. The purpose of this project is to study hormones in children. The investigators will look to see if a decrease of certain hormone levels affects how sick a child may become. This study is intended to develop a connection between hormone levels and severity of illness. It is hoped that the information gathered will help develop further studies that may more clearly explain the role of hormones in critically ill children and possibly the introduction of hormone replacement in critical illness.

DETAILED DESCRIPTION:
Neuroendocrine dysfunction is an abnormality in the production or release of certain hormones. Studies completed in adult patients have shown abnormal hormone levels in critical illness can contribute to how long patients stay in the intensive care unit, how severe their illness is and whether or not they survive. In children hormones are produced differently and have different functions. Depending on the particular illness in question hormonal dysfunction may have grave clinical consequences.

Thus far, there have been few studies that have examined neuroendocrine dysfunction in children. The aim of our study is to identify the common hormone responses in children, and to identify any connection between hormone levels and outcomes (likelihood of child staying in the intensive care unit for multiple days, etc.).

To explore these aims we will draw blood from all critically ill patients admitted to the pediatric intensive care unit (PICU) and check various hormone levels. Only those patients who require blood samples as part of their admission will have blood tests for certain hormone levels. No change will be made from established standard of care for a patient's particular critical illness.

The study is designed to examine hormone responses to critical illness and identify a connection between hormone levels and severity of illness. Based on these lab values we intend to lay a foundation for further studies that may more clearly explain the role of hormones in critically ill children, and possibly the introduction of hormone replacement in critical illness.

ELIGIBILITY:
Inclusion Criteria:

* All patients, birth - 18 years of age
* Admitted to the pediatric intensive care unit requiring blood to be drawn as part of medical management consistent with "standard of care".

Exclusion Criteria:

* Elective post-operative surgical patients.
* Pre-existing/known neuroendocrine disorder including, but not limited to, disorders of the hypothalamus, pituitary, adrenal, or thyroid gland.
* Patients being treated with or having a recent history of taking anti-psychotic medications (e.g. ingestion).
* Patients whose laboratory specimens have already been drawn prior to admission (emergency room or another facility) and who do not require further blood draws for medical management within a 12 hour window.

Min Age: 5 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients admitted to PICU
Sampling Method: Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2004-08; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
To determine the prevalence of neuroendocrine dysfunction in critically ill pediatric patients. | 13 months
  Conclued that neuroendocrine deficiency is present in critically ill pediatric patients. Prevalence is not greater in septic patients. Seventy-three children were enrolled over 13-month period. Larger scale studies are necessary to determine if presence of NEAD, or specific combinations of axis deficiency, is important in predicting outcomes or benefit of early hormonal replacement therapies in critically ill children.

CONTACTS AND LOCATIONS:
Overall Officials: James D Fortenberry, MD, Principal Investigator — Children's Healthcare of Atlanta
Locations (1):
- Children's Healthcare of Atlanta at Egleston, Atlanta, Georgia, United States